CLINICAL TRIAL: NCT04678830
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Leronlimab in Patients Experiencing Prolonged Coronavirus Disease 2019 (COVID-19) Symptoms [Long-Haulers]
Brief Title: Double Blind, Placebo Controlled Study of Safety and Efficacy of Leronlimab in Patients With "Long" COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD15_COVID-19
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Coronavirus Disease 2019
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — leronlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Syringes containing normal saline for injection were prepared by an unblinded pharmacist at the clinical sites for use as the placebo.
  Interventions: Drug: Placebos
- 700mg Leronlimab (Experimental): Each vial of active contains 350mg of leronlimab at a concentration of 175mg/ml (nominal 2mL fill volume) in formulation buffer containing histidine, glycine, sodium chloride, sorbitol, polysorbate 20 and sterile water for injections
  Interventions: Drug: Leronlimab (700mg)

INTERVENTIONS:
Drug: Placebos — Placebos
  Other Names: placebo
  Arms: Placebo
Drug: Leronlimab (700mg) — Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Other Names: Pro140
  Arms: 700mg Leronlimab

SUMMARY:
The purpose of this study is to assess the safety and efficacy of leronlimab (PRO 140) administered as weekly subcutaneous injections in subjects experiencing prolonged symptoms (> 12 weeks) of COVID-19.

DETAILED DESCRIPTION:
This is a Phase 2, two-arm, randomized, double blind, placebo controlled multicenter study to evaluate the safety and efficacy of leronlimab (PRO 140) in patients with prolonged symptoms caused by Coronavirus Disease 2019 (COVID-19). Patients will be randomized to receive weekly doses of 700 mg leronlimab (PRO 140), or placebo. Leronlimab (PRO 140) and placebo will be administered via subcutaneous injection.

The study will have three phases: Screening Period, Treatment Period, and Follow-Up Period. Total study duration is 91 days. The study will be conducted at up to 5 centers in the United States and planned number of subjects are 50 subjects.

Visit schedule:

Visit 1 - Screening assessment Visit 2 - baseline, first dose Visit 3 - no dose, baseline+3 days Visit 4 - second dose, baseline + 7 days Visit 5 - no dose, safety assessment/con med, baseline +10 days Visit 6 - third dose, baselines + 14 days Visit 7 - no dose, safety assessments, baseline + 17 days Visit 8 - fourth dose, baseline +21 days Visit 9 - no dose, safety assessment, baseline + 24 days Visit 10 - fifth dose, baseline + 28 days Visit 11 - no dose, safety assessment, baseline + 31 days Visit 12 - sixth dose, baseline + 35 days Visit 13 - no dose, safety assessment, baseline + 38 days Visit 14 - seventh dose, baseline + 42 days Visit 15 - no dose, safety assessment, baseline + 45 days Visit 16 - eighth and final dose, baseline + 49 days Visit 17 - End of treatment, baseline + 56 days

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult ≥ 18 years of age at time of enrollment.
2. Prior confirmed COVID-19 diagnosis by standard reverse transcriptase-polymerase chain reaction (RT-PCR) assay or equivalent testing
3. Clinical Symptom Score of ≥6 AND at least two symptoms of moderate or higher severity as listed below at the time of Screening and currently experiencing two or more of the following symptoms consistent with COVID-19 infection for a prolonged period of time (>12 weeks).

   Clinical symptoms include the following:
   * Respiratory symptoms such as cough, sore throat, stuffy or runny nose, shortness of breath (difficulty breathing), tightness of chest.
   * Neurological symptoms such as difficulty in concentration (brain fog), sleep disturbance/insomnia, headache, dizziness, anxiety, tingling or numbness, loss of sense of smell or taste.
   * Cardiovascular and Gastrointestinal symptoms such as feeling of fast heartbeat, nausea, vomiting, diarrhea.
   * Musculoskeletal symptoms such as muscle aches/cramps, muscle weakness, joint pain/swelling.
   * General immune response symptoms such as fatigue (low energy or tiredness), chills or shivering, feeling hot or feverish, or exertional malaise (feeling of discomfort, illness, or lack of well-being after physical activity or mental stress).

   Note: Clinical Symptom Score is obtained from the patient diary (refer to Appendix 1 for scoring instructions).
4. Electrocardiogram (ECG) with no clinically significant findings as assessed by the Investigator.

   Note: Below are the examples of clinically significant and non-clinically significant ECG abnormalities:
   * ECG findings indicative of acute myocardial infarction or acute ischemic changes would be considered clinically significant abnormalities.
   * ECG finding such as atrial fibrillation, atrial flutter, paced rhythms in individuals who have undergone permanent pacemaker placement, evidence of prior infarction, unchanged stable conduction abnormalities e.g. right bundle branch block, or any other finding which does not significantly impact mortality would be considered non-clinically significant findings and subjects with these abnormal findings would be allowed to enroll in the study.
5. Subject (or legally authorized representative) provides written informed consent prior to initiation of any study procedures.
6. Men and women of childbearing potential and their partner must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, bilateral tubal occlusion, or vasectomy) or must practice complete sexual abstinence for the duration of the study (excluding women who are not of childbearing potential and men who have been sterilized).
7. Females of child-bearing potential must have a negative urine pregnancy test at Screening Visit and prior to receiving the first dose of study drug; and Male participants must agree to use contraception and refrain from donating sperm for at least 90 days after the last dose of study intervention.
8. Subject is willing and able to comply with scheduled visits, drug administration plan, laboratory tests, other study procedures and study restrictions

Exclusion Criteria:

1. Exhibiting signs of moderate or severe pulmonary disease (such as Chronic Obstructive Pulmonary Disease (COPD), asthma, or pulmonary fibrosis)
2. Ongoing requirement of oxygen therapy
3. Pulse oxygen saturation (SpO2) of <94% on room air at the time of screening
4. History of splenectomy
5. Liver cirrhosis or patient showing signs of clinical jaundice at the time of screening
6. Chronic kidney disease stage 4 or requiring dialysis at the time of screening
7. New York Heart Association (NYHA) Class III or IV congestive heart failure (CHF)
8. Exhibiting signs of uncontrolled hypo-or hyper- thyroidism at the time of Screening
9. Uncontrolled rheumatologic disorders at the time of screening
10. History of organ transplantation or are candidates for organ transplantation at the time of screening
11. History of Chronic Fatigue Syndrome prior to COVID-19 infection
12. History of fibromyalgia prior to COVID-19 infection
13. History of major psychiatric disorder including bipolar disorders, schizophrenia, schizoaffective disorder, major depression. Patients with major depression can be enrolled if patient has had no episode within the past year or is considered in remission or controlled by treatment.
14. Any malignancy within the past 5 years, excluding successfully treated basal cell carcinoma or squamous cell carcinoma without evidence of metastases.
15. Any other clinically significant serious systemic diseases which would interfere with study conduct or study results interpretation per the Investigator.
16. Treatment with immunosuppressive or immunomodulatory medications within 5 half-lives prior to screening. Patients on replacement therapy for adrenal insufficiency will be allowed. Patients on stable (> 3 months) low dose corticosteroid ≤ 5 mg Prednisone will be allowed.
17. History of allergic reactions attributed to compounds of similar chemical or biologic composition to leronlimab (PRO 140) are not eligible
18. Ongoing use of CCR5 antagonist
19. Inability to provide informed consent or to comply with test requirements
20. Consideration by the investigator, for safety reasons, that the subject is an unsuitable candidate to receive study treatment
21. Pregnancy or breast feeding
22. Participating in another study for an investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2021-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Gaylis, MD, Principal Investigator — Arthritis and Rheumatic Disease Specialties Aventura Florida
Locations (2):
- United States (2):
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Center for Advanced Research & Education (CARE), Gainesville, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaylis NB, Ritter A, Kelly SA, Pourhassan NZ, Tiwary M, Sacha JB, Hansen SG, Recknor C, Yang OO. Reduced Cell Surface Levels of C-C Chemokine Receptor 5 and Immunosuppression in Long Coronavirus Disease 2019 Syndrome. Clin Infect Dis. 2022 Sep 30;75(7):1232-1234. doi: 10.1093/cid/ciac226. PMID 35452519
- [Derived] Chang XL, Wu HL, Webb GM, Tiwary M, Hughes C, Reed JS, Hwang J, Waytashek C, Boyle C, Pessoa C, Sylwester AW, Morrow D, Belica K, Fischer M, Kelly S, Pourhassan N, Bochart RM, Smedley J, Recknor CP, Hansen SG, Sacha JB. CCR5 Receptor Occupancy Analysis Reveals Increased Peripheral Blood CCR5+CD4+ T Cells Following Treatment With the Anti-CCR5 Antibody Leronlimab. Front Immunol. 2021 Nov 19;12:794638. doi: 10.3389/fimmu.2021.794638. eCollection 2021. PMID 34868084
- See also: PROMIS (Patient-Reported Outcomes Measurement Information System) Fatigue Assessment — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=66&Itemid=992
- See also: PROMIS (Patient-Reported Outcomes Measurement Information System) Cognitive Function Assessment — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=748&Itemid=992
- See also: PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance Assessment guide — https://www.healthmeasures.net/index.php?option=com_instruments&view=measure&id=70&Itemid=992
- See also: PROMIS T-score maps — https://www.healthmeasures.net/score-and-interpret/interpret-scores/promis/t-score-maps

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty six (56) subjects were enrolled in the study with 28 subjects in each treatment arm. All patients were enrolled under protocol version 3.0 (effective date 25-Feb-2021). The study was performed between 01 March 2021 and 01 July 2021.
Period: Overall Study
Arm/Group | Placebo | 700mg Leronlimab
Started | 28 | 28
Completed | 26 | 27
Not Completed | 2 | 1
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Modified Intent-to-Treat (mITT) population is defined as the set of subjects who have received at least one dose of study treatment (leronlimab or placebo). This population was used for the analysis of efficacy parameters or measurements.
  The Safety Population includes all subjects who received one dose of study treatment (leronlimab or placebo). This population was used for the analysis of safety parameters or measurements.
Groups:
- Total: Total of all reporting groups
Arm/Group | 700mg Leronlimab | Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.8) | 51.6 (13.2) | 48.6 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56
Baseline COVID-19 Related Symptom Score [Mean (Standard Deviation); unit: units on a scale] | 32.5 (9.96) | 26.9 (10.19) | 29.4 (10.64)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Daily COVID-19-related Symptom Severity Score Through Day 56.
Description: Changes in common COVID-19-related symptoms were evaluated daily by the patient using a patient diary between start and end of treatment. The diary is shown in Appendix 17.1 in the protocol and covers patient-reported changes for symptoms (ranked as none = 0, mild = 1, moderate = 2 or severe = 3) of cough, sore throat, stuffy or runny nose, difficulty breathing, feeling tightness in chest, feeling fast heartbeat, fatigue, exertional malaise, muscle aches and cramps, muscle weakness, joint pain and swelling, shivering and chills, feeling hot or feverish, difficulty concentrating, insomnia, headache, dizziness, anxiety, tingling or numbness, nausea, vomiting, diarrhea, sense of smell, sense of taste. Maximum score could be 70 (22 parameters with scores up to 3, two parameters with scores up to 2), lowest score could be 0. A negative value shows improvement in symptoms. The lower the value, the greater the improvement (i.e., a score of -16 is greater improvement than a score of -8).
Time Frame: Changes in COVID-19 related symptoms from baseline (start of treatment) and day 56 (end of treatment)
Population: The Modified Intent-to-Treat (mITT) population was defined as the set of subjects who received at least one dose of leronlimab (PRO 140) or placebo. This population was to be used for the analysis of efficacy parameters or measurements. Fifty six (56) patients received at least one dose of leronlimab or placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale | -16.3 (13.14) | -8.1 (12.27)

2. Secondary Outcome: Duration of COVID-19 Associated Symptoms From Start of Study Treatment (Day 0) Based on Self-assessment Using Daily Symptom Diary.
Description: Number of days when any symptoms scored as moderate or severe at baseline (Day 0) are still scored as moderate or severe through day 56 (end of treatment) or symptoms scored as mild or absent at baseline are scored as mild or worse at day 56 (end of treatment).
Time Frame: Duration of symptoms from baseline (day 0, start of treatment) and day 56 (end of treatment)
Population: mITT
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
days
  Duration (days) of cough | 14.9 (18.8) | 7.8 (12.8)
  Duration (days) of sore throat | 10.6 (15.7) | 9.4 (13.4)
  Duration (days) of Stuff/Runny Nose | 19.3 (23.0) | 20.7 (20.9)
  Duration (days) of shortness of breath | 11.5 (17.4) | 13.9 (17.4)
  Duration (days) of tightness of chest | 10.3 (14.8) | 12.3 (17.1)
  Duration (days) of fast heartbeat | 14.8 (18.7) | 16.0 (15.6)
  Duration (days) of fatigue | 6.5 (14.0) | 10.6 (18.4)
  Duration (days) of exertional malaise | 12.7 (18.8) | 10.6 (15.3)
  Duration (days) muscle aches / cramps | 16.5 (19.6) | 17.7 (16.6)
  Duration (days) of Muscle Weakness | 17.1 (19.4) | 20.8 (17.9)
  Duration (days) joint pain/swelling | 15.9 (16.7) | 18.3 (18.6)
  Duration (days) of chills or shivering | 6.6 (11.1) | 3.9 (7.7)
  Duration (days) of feeling hot or feverish | 10.5 (13.6) | 9.9 (16.2)
  Duration (days) of difficulty in concentration | 15.6 (20.3) | 11.8 (17.7)
  Duration (days) of sleep disturbance | 13.3 (17.2) | 14.4 (17.5)
  Duration (days) of headache | 16.0 (16.6) | 17.8 (18.0)
  Duration (days) of dizziness | 11.8 (17.6) | 16.9 (18.6)
  Duration (days) of anxiety | 16.8 (22.3) | 15.1 (17.4)
  Duration (days) of tingling or numbness | 14.0 (19.3) | 18.3 (19.4)
  Duration (days) of nausea | 6.8 (9.8) | 8.5 (12.5)
  Duration (days) of vomiting | 0.3 (0.7) | 0.6 (1.6)
  Duration (days) of diarrhea | 8.5 (13.7) | 7.1 (9.5)
  Duration (days) of change to sense of smell | 16.8 (21.2) | 8.5 (15.5)
  Duration (days) in change of sense of taste | 13.5 (18.3) | 8.6 (17.0)

3. Secondary Outcome: Number of Days Free of Symptoms Associated With COVID-19 That Were Present at the Start of Study Treatment (Day 0) Based on Self-assessment Using Daily Symptom Diary.
Description: Symptom-free days are defined as number of days when any symptoms scored as mild, moderate or severe at baseline are scored as absent (or none) through Day 56 (end of treatment) using a self-assessment diary.
Time Frame: Between start of treatment (day0) and day 56 (end of treatment)
Population: mITT
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
Days
  Days free of cough | 16.8 (19.4) | 11.3 (17.1)
  Days free of sore throat | 4.9 (9.8) | 11.5 (18.5)
  Days free of stuffy or runny nose | 8.7 (13.2) | 12.8 (17.7)
  Days free of shortness of breath | 8.2 (12.0) | 15.0 (17.0)
  Days free of tightness of chest | 10.3 (16.1) | 13.4 (19.0)
  Days free of fast heartbeat | 12.8 (16.5) | 16.4 (18.8)
  Days free of fatigue | 3.9 (7.5) | 5.4 (10.9)
  Days free of exertional malaise | 7.2 (10.5) | 11.1 (15.0)
  Days free of muscle aches and cramps | 9.1 (13.7) | 14.2 (15.5)
  Days free of muscle weakness | 9.5 (14.7) | 12.0 (16.1)
  Days free of joint pain/swelling | 10.5 (17.8) | 5.1 (12.7)
  Days free of chills or shivering | 12.6 (19.4) | 16.6 (21.6)
  Days free of being hot or feverish | 14.8 (20.4) | 14.5 (18.2)
  Days free from difficulty concentrating | 4.6 (9.1) | 7.4 (13.3)
  Days free from sleep disturbance | 10.3 (12.1) | 13.6 (15.7)
  Days free from headache | 15.4 (16.2) | 12.5 (16.4)
  Days free from dizziness | 11.0 (18.5) | 9.9 (15.3)
  Days free from anxiety | 5.1 (11.0) | 12.4 (16.4)
  Days free from tingling or numbness | 16.5 (20.1) | 9.0 (15.8)
  Days free from nausea | 14.0 (19.8) | 13.9 (18.1)
  Days free from diarrhea | 8.3 (15.0) | 13.6 (18.3)
  Days free from change in sense of smell | 7.8 (14.2) | 6.9 (15.3)
  Days free from change in sense of taste | 8.8 (16.3) | 8.0 (16.9)

4. Secondary Outcome: Progression (or Worsening) of COVID-19-associated Symptoms Through Day 56 Compared to Baseline.
Description: Progression or worsening of symptoms is defined as number of days when any symptoms scored as 2 at baseline scored as 3 through day 56 or 1 at baseline are scored as 2 or 3 through day 56 or scored 0 at study entry scored as 1, 2 or 3 through day 56. No change in symptoms would give a score of 0, symptom progression would give a positive number, symptom improvement would a negative number. Minimum baseline symptom score for eligibility for the study was 6. Maximum symptom score is 70, therefore if all symptoms progressed to the severest level the change in score would be +64. If all patients had a severe score for all symptoms at baseline and all improved to no symptoms at day 56, the maximum improvement in score would be -70.
Time Frame: Between start of treatment (day0) and day 56 (end of treatment)
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 23 | 25
score on a scale
  Cough | -0.6 (0.8) | -0.4 (0.9)
  Sore throat | -0.1 (0.7) | -0.2 (0.8)
  Stuffy or runny nose | -0.7 (0.8) | -0.1 (0.8)
  Shortness of breath | -0.8 (1.0) | -0.6 (0.9)
  Tightness of chest | -0.6 (0.9) | -0.3 (0.9)
  Fast heartbeat | -0.8 (0.8) | -0.5 (1.0)
  Fatigue | -1.1 (0.9) | -1.1 (1.0)
  Exertional Malaise | -1.1 (1.1) | -0.9 (1.0)
  Muscle aches and cramps | -0.9 (0.9) | -0.7 (0.9)
  Muscle weakness | -0.9 (1.1) | -0.5 (0.8)
  Joint Pain/swelling | -0.8 (0.7) | -0.3 (0.9)
  Chills and shivering | -0.6 (0.6) | -0.5 (0.8)
  Hot or feverish | -0.5 (0.8) | -0.6 (1.1)
  Difficulty in concentrating | -1.0 (1.0) | -1.1 (1.0)
  Sleep disturbance | -1.2 (0.9) | -1.1 (1.0)
  Headache | -1.0 (1.0) | -0.7 (1.0)
  Dizziness | -0.7 (1.0) | -0.4 (0.9)
  Anxiety | -0.7 (0.9) | -0.8 (0.8)
  Tingling or numbness | -0.8 (1.0) | -0.3 (0.9)
  Nausea | -0.6 (0.9) | -0.5 (0.9)
  Vomiting | 0.0 (0.1) | 0.0 (0.1)
  Diarrhea | -0.0 (0.6) | -0.6 (1.0)
  Sense of Smell | -0.3 (0.5) | -0.2 (0.4)
  Sense of taste | -0.3 (0.5) | -0.2 (0.4)

5. Secondary Outcome: Change From Baseline in PROMIS® Fatigue Score at Days 7,14, 21, 28, 35, 42 and End of Treatment (Day 56).
Description: Change from baseline in physical and psychological fatigue measured using the PROMIS® scale. A decrease in the score compared to baseline shows an improvement in the symptom. PROMIS definition - Patient-Reported Outcomes Measurement Information System. The Fatigue Short Form (4a) was used (Section 17.3 Appendix 3 of protocol). Raw fatigue scores range from 4 to 20 and are converted to a T-score metric where the response from the general population is set at 50 with standard deviations at 10; a score of greater than 60 would be one std dev greater than the general population, meaning more fatigue. A link to the fatigue score maps is provided in the hyperlinks section. The minimum fatigue T-score is 33.7 (with a std error of 4.9) and a maximum score of 75.8 (with a std error of 3.9). The higher the score, the more fatigue. A decrease in the fatigue score from baseline to day 28 and day 56 would indicate decrease in fatigue.
Time Frame: Between Baseline (day 0), Visit 4 (day 7), Visit 6 (day 14), Visit 8 (day 21) Visit 10 (day 28), Visit 12 (day 35), Visit 14 (day 42), Visit 16 (Day 56) and Visit 17 (day 56, end of treatment).
Population: mITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
Units on a scale
  Baseline score (day 0) | 68.4 (6.5) | 66.6 (7.1)
  Change from baseline to visit 4 (day 7) | -5.3 (9.9) | -6.1 (8.5)
  Change from baseline to visit 6 (day 14) | -7.6 (10.7) | -7.6 (8.5)
  Change from baseline to visit 8 (day 21) | -8.4 (14.6) | -10.2 (10.1)
  Change from baseline to visit 10 (day 28) | -8.8 (12.1) | -7.5 (10.5)
  Change from baseline to Visit 12 (day 25) | -11.1 (13.4) | -8.6 (10.8)
  Change from baseline to visit 14 (day 42) | -11.0 (14.0) | -8.1 (11.2)
  change from baseline to visit 16 (day 49) | -11.8 (12.9) | -11.0 (11.5)
  Change from baseline to end of treatment (day 56) | -11.1 (11.9) | -10.2 (10.8)

6. Secondary Outcome: Change From Baseline in PROMIS® Cognitive Function Score at Days 7, 14, 21, 28, 35, 42, 49 and End of Treatment (d56)
Description: Change in cognitive function score between baseline, day 28 and day 56 were measured using the PROMIS Cognitive Function Assessment Short Form 4a. Higher scores on the PROMIS Cognitive Function Assessment indicate better perceived cognitive functioning. Answers to 4 questions with scores ranging from 1 (very often - several times a day) to 5 (never) provide raw scores that are then normalized T scores. A T score of 50 is the mean of the general population, with std devs of 10, therefore a score of 40 is one std dev lower than that of the general population. The lowest raw score (4) converts to a T score of 24.99 while the highest raw score (20) converts to a T score of 61.13. A link to the PROMIS scoring maps is provided in the hyperlinks section. An increase in score for cognitive function assessment represents an increase in cognitive function
Time Frame: Baseline (start of treatment), day 28 and day 56 (end of treatment)
Population: mITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
units on a scale
  Baseline (day 0) | 29.6 (5.5) | 34.6 (9.5)
  Change from baseline to visit 4 (day 7) | 5.1 (8.9) | 2.7 (8.2)
  Change from baseline to visit 6 (day 14) | 7.4 (9.6) | 4.9 (9.5)
  Change from baseline to visit 8 (day 21) | 7.4 (10.0) | 4.6 (7.9)
  Change from baseline to visit 10 (day 28) | 9.0 (8.9) | 4.1 (8.0)
  Change from baseline to visit 12 (day 35) | 10.1 (9.4) | 6.2 (9.1)
  Change from baseline to visit 14 (day 42) | 10.8 (11.2) | 6.2 (8.6)
  Change from baseline to visit 16 (day 49) | 10.3 (10.8) | 7.4 (9.7)
  Change from baseline to end of treatment (day 56) | 10.9 (10.8) | 6.3 (8.8)

7. Secondary Outcome: Change From Baseline in PROMIS® Sleep Disturbance Score at Days 7,14, 21, 28, 35, 42, 49 and End of Treatment (Day 56).
Description: Assessment of change in sleep disturbance between baseline, day 28 and day 56 used the PROMIS® Sleep Disturbance Short Form (see Appendix 5 in Section 17 of the protocol). Four questions are scored between 1 (best score for good quality sleep) and 5 (worst score) such that the lower the score, the better the sleep. Raw scores are converted to a T-score with a mean of 50 and a standard deviation (SD) of 10 for the general population. T-scores of 60 are one SD worse than average (worse quality sleep). By comparison, Sleep Disturbance T-scores of 40 are one SD better than average. The PROMIS Sleep Disturbance scoring manual shows the lowest sleep disturbance score of 4 converting to a T score of 32 with a std error of 5.2, while the highest score of 20 converts to a T score of 73.3 with a std error of 4.6. The change from baseline is based on patients with paired values.
Time Frame: as for outcome 5
Population: mITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
score on a scale
  Baseline score (day 0) | 60.2 (8.0) | 58.3 (8.5)
  Change from baseline to visit 4 (day 7) | -4.1 (8.6) | -1.9 (6.2)
  Change from baseline to visit 6 (day 14) | -5.3 (9.6) | -3.4 (8.0)
  Change from baseline visit 8 (day 21) | -7.7 (10.2) | -5.1 (7.1)
  Change from baseline to visit 10 (day 28) | -7.2 (8.9) | -5.7 (9.2)
  Change from baseline to visit 12 (day 35) | -8.3 (10.8) | -4.2 (6.5)
  Change from baseline to visit 14 (day 42) | -7.7 (10.7) | -5.3 (7.9)
  Change from baseline to visit 16 (day 49) | -7.6 (9.5) | -6.0 (10.4)
  Change from baseline to end of treatment (day 56) | -8.3 (9.4) | -5.5 (9.4)

8. Secondary Outcome: Number of Participants Requiring Hospitalization During the Treatment Phase
Description: Number of participants who required hospitalization during the treatment phase.
Time Frame: Between baseline (start of treatment) and day 56 (end of treatment)
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
Participants | 0 | 0

9. Secondary Outcome: Duration (Days) of Hospitalization During the Treatment Phase
Description: Duration (in days) of hospitalization required during treatment phase
Time Frame: Between baseline (start of treatment) and day 56 (end of treatment)
Population: mITT
Measure: Number; unit: days
Arm/Group | 700mg Leronlimab | Placebo
Number analyzed (Participants) | 28 | 28
days | 0 | 0

10. Other Pre Specified Outcome: Change From Baseline in Pulse Oxygen Saturation (SpO2) at Day 7, 14, 21, 28, 35, 42, 49, and 56
Description: Exploratory Outcome - Change from baseline in pulse oxygen saturation (SpO2) at Day 7, 14, 21, 28, 35, 42, 49, and 56
Time Frame: Change between baseline (start of treatment) and Day 7, 14, 21, 28, 35, 42, 49, and 56 (end of treatment).
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change From Baseline in Serum Cytokine and Chemokine Levels on Days 28 and 56.
Description: Exploratory Outcome - Change from baseline in serum cytokine and chemokine levels
Time Frame: Change between baseline (start of treatment) and days 28 and 56 (end of treatment)
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change From Baseline in CD4+ and CD8+ T Cell Count on Days 28 and 56.
Description: Exploratory Outcome - Change from baseline in CD4+ and CD8+ T cell count
Time Frame: Change between baseline (start of treatment) and days 28 and 56 (end of treatment)
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline in Transforming Growth Factor Beta 1 (TGF beta1) on Days 28 and 56
Description: Exploratory Outcome - change in TGF-b1 from baseline to days 28 and 56 (end of treatment)
Time Frame: Change between baseline (start of treatment) and days 28 and 56 (end of treatment)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change From Baseline in C-reactive Protein (CRP) on Days 28 and 56
Description: Exploratory Outcome - Change in C-reactive Protein (CRP) from baseline to Days 28 and 56 (end of treatment)
Time Frame: Change between baseline (start of treatment) and days 28 and 56 (end of treatment)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change From Baseline in CCR5 Receptor Occupancy on Days 28 and 56.
Description: Exploratory Outcome - Change in CCR5 receptor occupancy from baseline and days 28 and 56 (end of treatment)
Time Frame: Change between baseline (start of treatment) and days 28 and 56 (end of treatment)
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploration of Biomarkers That May Predict and/or Act as Pharmacodynamic Indicators of Pharmacologic Activity of Leronlimab.
Description: Exploratory Outcome - Exploration of biomarkers that may predict and/or act as pharmacodynamic indicators of pharmacologic activity of leronlimab.
Time Frame: 91 Days
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Incidence of Treatment-related Adverse Events (TEAEs)
Description: Safety Measurement - incidence of treatment emergent adverse events
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Incidence and Severity of Treatment-emergent Adverse Events (TEAEs)
Description: Safety Measures - Incidence and severity of treatment-emergent adverse events
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Incidence of Serious Adverse Events (SAEs)
Description: Safety Measures - incidence of severe adverse events
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Incidence of TEAEs and SAEs Leading to Discontinuation of Study Medication.
Description: Safety Measures - incidence of TEAEs and SAEs leading to discontinuation of study medication
Time Frame: Between baseline and day 56
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Changes in Blood Chemistry, Hematology and Coagulation Parameter Results
Description: Safety Measures - Changes in blood chemistry, hematology and coagulation parameter results
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Changes in Vital Signs Including Temperature, Pulse, Respiratory Rate, Systolic and Diastolic Blood Pressure
Description: Safety Measures - Changes in vital signs including temperature, pulse, respiratory rate, systolic and diastolic blood pressure
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Changes in Physical Examination Results
Description: Safety Measures - Changes in physical examination results
Time Frame: Between baseline and day 91
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Changes in Electrocardiogram (ECG) Results
Description: Safety Measures - changes in electrocardiogram results
Time Frame: Change between baseline and day 91
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected between start of treatment (baseline, day 0) and 28 days after end of treatment. First dose was administered on Day 0, last dose (dose 8) was administered on day 49, End of Treatment (EOT) was 7 days after last dose (day 56) and follow-up was for the 28 day period after the EOT visit.
Arm/Group | 700mg Leronlimab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/28
Other Adverse Events (participants affected / at risk) | 22/28 | 20/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 700mg Leronlimab (N=28) | Placebo (N=28)
Seizures and seizure disorders (Nervous system disorders) | 0 (0) | 1 (1) — Worsening seizures
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 700mg Leronlimab (N=28) | Placebo (N=28)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diaphragmatic Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Swollen Tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site pruritis (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 2 (2) | 0 (0) — General disorders and injection site reaction
Malaise (General disorders) | 2 (2) | 0 (0) — General Disorders and Injection Site Reactions
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Bacterial Vaginosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal Infection (Infections and infestations) | 2 (2) | 2 (2)
Fungal Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 2 (2)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hyperreflexia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaethesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis - contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Keratomileusis (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Blue toe syndrome (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT04678830/Prot_SAP_ICF_001.pdf